CLINICAL TRIAL: NCT02404038
Title: An Open-Label, Randomized Crossover Study to Evaluate the Acceptability and Preference for Contraceptive Options in Healthy HIV-Uninfected Female Adolescents, 16-17 Years of Age, as Proxy for HIV Prevention Methods
Brief Title: A Study to Evaluate the Acceptability and Preference for Contraceptive Options as Proxy for HIV Prevention Methods
Acronym: UChoose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Desmond Tutu HIV Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Protocol A: UChoose
Record Dates: First submitted 2015-03-10; First posted 2015-03-31 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: HIV
Keywords: choice; young women; adolescent girls; preference
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Injectable (Active Comparator): This arm will receive Nur-Isterate administered as an intramuscular injection administered bi-monthly (every 8 weeks).
  Interventions: Drug: Nur-Isterate
- Arm B: Intra-vaginal (Active Comparator): This arm will receive the Nuvaring a combined hormonal contraceptive intravaginal ring, inserted once every 28 days, and removed after 21 days.
  Interventions: Device: Nuvaring
- Arm C: Oral (Active Comparator): This arm will receive Triphasil a daily oral contraceptive of 21 active tablets followed by 7 inert tablets, starting initially on first day of menstrual cycle
  Interventions: Drug: Triphasil

INTERVENTIONS:
Drug: Nur-Isterate — Nur-Isterate is a progestogen-only injectable contraceptive (POIC) is a long-acting, reversible contraceptive. Nur-Isterate is administered as an intramuscular injection administered bi-monthly (every 8 weeks). Each ampoule of Nur-Isterate contains 1ml/200mg of norethisterone enantate (17alpha-ethinyl-17beta-heptanoyloxy-4-estrene-3-one).
  Arms: Arm A: Injectable
Device: Nuvaring — Nuvaring is the trade name for a combined hormonal contraceptive intravaginal ring, inserted once every 28 days, and removed after 21 days. The flexible plastic ring works in a similar way to the oral contraceptive pill to prevent pregnancy. It contains etonogestrel/ethinyl estradion and delivers 0.120mg/0.015mg per day.
  Arms: Arm B: Intra-vaginal
Drug: Triphasil — Triphasil is a daily oral contraceptive: 21 active tablets followed by 7 inert tablets, starting initially on first day of menstrual cycle
  Composition:
  The six brown tablets of TRIPHASIL contain 30 µg ethinyl oestradiol and 50 µg levonorgestrel.
  The five white tablets contain 40 µg ethinyl oestradiol and 75 µg levonorgestrel.
  The ten yellow tablets contain 30 µg ethinyl oestradiol and 125 µg levonorgestrel.
  The seven red tablets are inert
  Arms: Arm C: Oral

SUMMARY:
This study will enrol sexually active, healthy girls aged 16-17 to assess and compare the acceptability and preference for a monthly vaginal ring, bi-monthly injectable contraception or daily dose oral contraception, as proxy for female-controlled ARV-based HIV prevention methods.

DETAILED DESCRIPTION:
The family planning field has shown the importance of providing sufficient choice to meet individuals' changing needs and preferences, and has demonstrated that diversifying delivery modes and dosing options is key to expanding acceptability, use and continuation of contraceptive products. It is not yet clear to what extent choice and preference of modes of delivery will play in the biomedical HIV prevention world. It may be possible that closely associated with the behavioural components of decision to use, uptake, and consistent adherence to prevention products will hinge on a sense that a particular modality is preferred or suits an individual compared to other modalities. Vaginal rings, pills, and injectables have already proven successful in the field of contraception, and therefore may act as surrogates for a range of HIV prevention delivery options that may help to meet the different sexual and reproductive health concerns of women.

A better understanding of the population of adolescents seeking contraception can also help researchers understand the acceptability and feasibility of, as well as adherence to similar modes of delivery for HIV prevention options. By using contraceptive methods as a proxy for available female-controlled HIV prevention delivery methods, such as microbicides and PrEP, we propose to examine in detail, the acceptability of these surrogates to adolescent women; their preferences for mode of delivery; and their adherence barriers and facilitators thereof to such products. Three contraceptive options will be used in this study to emulate the modes of delivery currently being developed for HIV prevention options: (1) monthly vaginal ring (NuvaRing), (2) bi-monthly injectable contraception (Nuristerate) and (3) daily dose oral contraception (Triphasil or Nordette).

This is an open-label, randomized crossover study of 150 sexually active female adolescents (>16 and <18 years) to be recruited, with parental consent, and randomly assigned to a monthly vaginal ring, bi-monthly injectable contraception, or daily dose oral contraception at baseline. After 4 months, participants will crossover, ensuring that all participants use the vaginal ring, and either the oral contraceptive or the bi-monthly injectable contraceptive throughout the course of the study. Participants will be followed for a total of 8 months.

Upon enrollment participants will be randomly assigned in a 1:1:1 ratio to one of three study arms (50 participants per arm):

Arm 1/Group A: Participants will receive an injectable contraceptive once every 8 weeks for a 4 month period.

Arm 2/Group B: Participants will receive the contraceptive intravaginal NuvaRing to be inserted once every 28 days (and removed after 21 days of each 28 day insertion) for a 4 month period

Arm 3/Group C: Participants will be supplied with oral contraceptives and will be required to take a daily tablet for 21 days each month and a placebo tablet for days 22 to 28 each month, for a 4 month period.

After 4 months, participants in Group A and Group C will be assigned to Group B; participants in Group B will be allowed to select either Groups A or Group C, ensuring that all participants use the vaginal ring, and most either the oral contraceptive or the bi-monthly injectable contraceptive.

Participants will attend follow-up visits every 8 weeks throughout the duration of the study. Those participants receiving the oral contraceptive or intravaginal ring will therefore receive 8 weeks' product supply at each visit. At each visit preference / acceptability, sexual behaviour and adherence to study product will be assessed using mainly quantitative measures and general attitudes and experiences of use will be assessed in focus group discussions at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 to 17 years (inclusive) at screening, verified per study site SOPs.
2. Able and willing to provide written informed consent and has a guardian who is able and willing to provide written informed consent to be screened for and to take part in the study.
3. Report being sexually active, as defined by penetrative vaginal sex in the last 90 days.
4. (For those potential participants who are currently using a method of hormonal contraception) Reports being within 30 days or less of needing a new supply of contraception; agrees to terminate her current method of contraception; and indicates willingness to use the contraceptive options as assigned in the study.
5. Able and willing to provide adequate locator information, as defined in site SOPs.
6. HIV-uninfected based on testing performed by study staff at screening and enrollment.
7. Has negative pregnancy test at screening and enrollment and per participant report, does not intend to become pregnant in the next 8 months.
8. Agrees to use condoms, in addition to the assigned contraception options, for the duration of the study
9. Does not report intention to relocate out of the study area during the course of the study.
10. At Screening/ Enrollment, participant states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina, including but not limited to, spermicides, diaphragms, contraceptive vaginal rings (besides the Nuvaring), vaginal medications, menstrual cups, cervical caps (or any other vaginal barrier method), douches, lubricants, sex toys (vibrators, dildos, etc) throughout the duration of study participation.
11. Does not have job or other obligations that would require long absences from the area (> 8 weeks at a time).
12. Willing to undergo all study-required procedures.
13. At screening and enrollment, agrees not to participate in other research studies involving medical devices or vaginal products for the next 32 weeks

Exclusion Criteria:

1. Diagnosed with pelvic inflammatory disease, a sexually transmitted infection (STI) or reproductive tract infection (RTI) requiring treatment per current WHO guidelines.

   Note: Otherwise eligible participants diagnosed with STI or RTI during screening will be offered treatment and may be enrolled after completing treatment and all symptoms have resolved.
2. Urine dipstick for protein and glucose, of more than > 1+.
3. Any Grade > 2 toxicity on screening tests and assessments.
4. Has any other condition that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.
5. Known allergy or sensitivity to the study products.
6. Demonstrates intent or desire to conceive in the next 32 weeks.
7. Appears psychologically unstable, intoxicated or under the influence of alcohol or other drugs at the time of informed consent.
8. Has any other condition that, in the opinion of the investigator/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
9. Has hormonal contraceptive implant device or an intrauterine contraceptive device.

Ages: 16 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07-14 (Actual); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
13-item Ortho Birth Control satisfaction assessment tool to measure acceptability of each contraceptive option | 32 weeks
  questionnaire administered after every 8 weeks on each contraceptive method

SECONDARY OUTCOMES:
self-report, returned pill packs and rings to measure adherence to each contraceptive method | 8 weeks, 16 weeks, 24 weeks & 32 weeks
  interviewer-administered questionnaire on adherence to product, pill counts and visual inspection of rings
self-reported measure of the impact of contraceptive method use on sexual risk behavior | baseline, 8 weeks, 16 weeks, 24 weeks & 32 weeks
  interviewer-administered questionnaires measuring sexual risky behavior, ie. number of sexual partners, condom use, alcohol use
qualitative measures of perceptions on key issues associated with each method of contraceptive measured in focus group discussions | 8 months
  in-depth interviews and focus group discussions with participants who used the products

OTHER OUTCOMES:
through self-reports and interviewer-administered questionnaires explore how perceptions may be extrapolated to ART based HIV prevention methods | 8 months
  self-administered measure of HIV prevention preferences, ORTHO Birth Control satisfaction measure tool

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, MBChB, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Desmond Tutu HIV Centre, Cape Town, South Africa

REFERENCES:
- [Derived] Fynn L, Gill K, Wallace M, Atujuna M, Duyver M, Ngcobo P, Spiegel H, Rinehart A, Hosek S, Bekker LG. "It's already in your body and it's preventing": a qualitative study of African female adolescent's acceptability and preferences for proxy HIV prevention methods in Cape Town, South Africa. BMC Public Health. 2023 Nov 2;23(1):2143. doi: 10.1186/s12889-023-16955-3. PMID 37919697
- [Derived] Happel AU, Gasper M, Balle C, Konstantinus I, Gamieldien H, Dabee S, Gill K, Bekker LG, Passmore JS, Jaspan HB. Persistent, Asymptomatic Colonization with Candida is Associated with Elevated Frequencies of Highly Activated Cervical Th17-Like Cells and Related Cytokines in the Reproductive Tract of South African Adolescents. Microbiol Spectr. 2022 Apr 27;10(2):e0162621. doi: 10.1128/spectrum.01626-21. Epub 2022 Mar 29. PMID 35348351
- [Derived] Balle C, Konstantinus IN, Jaumdally SZ, Havyarimana E, Lennard K, Esra R, Barnabas SL, Happel AU, Moodie Z, Gill K, Pidwell T, Karaoz U, Brodie E, Maseko V, Gamieldien H, Bosinger SE, Myer L, Bekker LG, Passmore JS, Jaspan HB. Hormonal contraception alters vaginal microbiota and cytokines in South African adolescents in a randomized trial. Nat Commun. 2020 Nov 4;11(1):5578. doi: 10.1038/s41467-020-19382-9. PMID 33149114
- [Derived] Gill K, Happel AU, Pidwell T, Mendelsohn A, Duyver M, Johnson L, Meyer L, Slack C, Strode A, Mendel E, Fynn L, Wallace M, Spiegel H, Jaspan H, Passmore JA, Hosek S, Smit D, Rinehart A, Bekker LG. An open-label, randomized crossover study to evaluate the acceptability and preference for contraceptive options in female adolescents, 15 to 19 years of age in Cape Town, as a proxy for HIV prevention methods (UChoose). J Int AIDS Soc. 2020 Oct;23(10):e25626. doi: 10.1002/jia2.25626. PMID 33034421
- [Derived] Balle C, Gill K, Konstantinus IN, Jaumdally SZ, Lennard K, Esra R, Happel AU, Barnabas SL, Gamieldien H, Pidwell T, Maseko V, Lesosky M, Myer L, Passmore JS, Bekker LG, Jaspan HB. Hormonal contraception and risk of STIs and bacterial vaginosis in South African adolescents: secondary analysis of a randomised trial. Sex Transm Infect. 2021 Mar;97(2):112-117. doi: 10.1136/sextrans-2020-054483. Epub 2020 Sep 28. PMID 32989170